CLINICAL TRIAL: NCT05347511
Title: Study of the Pronostic Impact of Immunohistochemical, Histological, Radiological and Molecular Factors in Patients With Primary Central Nervous System Lymphoma
Brief Title: Study of the Pronostic Impact of Immunohistochemical, Histological and Radiological Factors in Patients With Primary Central Nervous System Lymphoma.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Guillaume GAUCHOTTE, PUPH, Central Hospital, Nancy, France
Other Study IDs: 2022PI003
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Rare Disease With Poor Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Adults' immunocompetent patients treated at the University Hospital of Nancy are included if they had a DLBCL's PCNSL diagnosed between January 2011 and December 2019, without regard to the clinical outcome.. All the patients are included in the LOC network database (Lymphomes oculo-cerebraux) and had given their written consent for the use of their samples for studies. Biological and clinical data will be collected for each patient from original medical charts.
  Formalin-fixed paraffin-embedded (FFPE) are available for 90 patients and will be used for NGS and Immunohistochemistry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary Central Nervous System Lymphoma (PCNSL) have a specific mutational profile in comparison to systemic diffuse large cells lymphoma (DLBCLs) that can be related to the expression of immunohistochemical markers as cyclon, NPM1, CD30, and P53 which could be predictive factor for prognosis and/or chemotherapy response. The main objective of this study is to identify new prognostic factors and new potential therapeutic targets.

The secondary objectives are to correlate the histological, the radiological and the clinical's informations of these patients.

ELIGIBILITY:
Inclusion Criteria:

* PCNSL diagnosed between January 2011 and December 2019, without regard to the clinical outcome.
* Age > 18

Exclusion Criteria:

* Systemic DLBCL

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults' immunocompetent patients treated at the University Hospital of Nancy are included if they had a DLBCL's PCNSL diagnosed between January 2011 and December 2019, without regard to the clinical outcome.. All the patients are included in the LOC network database (Lymphomes oculo-cerebraux) and had given their written consent for the use of their samples for studies. Biological and clinical data will be collected for each patient from original medical charts.
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2022-04-20 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
correlation between the survival and the expression of Cyclon, NPM1 and CD30. | 17/10/2022
  kaplan meyer

SECONDARY OUTCOMES:
the correlation between the molecular abnormalities and the expression of Cyclon, NPM1 and CD30 | 17/10/2022
  mutational signature

IPD SHARING:
Plan to Share IPD: No